CLINICAL TRIAL: NCT06357273
Title: White Tea Consumption Alleviates on Body Composition, Oxidative Stress, Appetite Hormones, Inflammation and Lipids in Obese Patients
Brief Title: The Effect of White Tea Consumption on Obesity
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Kerimali Akyıldız, Lecturer, Recep Tayyip Erdogan University
Other Study IDs: WhiteTeaAY
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Obesity; Obesity; Endocrine; Obesity Adult Onset
Keywords: White tea; Obesity; Weight loss; Appetite hormones; Inflammation; Lipid profile
MeSH Terms: conditions — Obesity; Weight Loss; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples obtained from routine laboratory investigations were retrieved (10 mL). Serum glucose, total cholesterol, low density lipoprotein cholesterol, high density lipoprotein cholesterol and triglyceride were determined with an autoanalyzer. Human-specific ELISA kits were used to measure leptin, adiponectin, ghrelin, asprosin, tumor necrosis factor alpha, interleukin- 6, interleukin-1β, matrix metallopeptidase-9, pancreatic lipase and 8-hydroxy-2' -deoxyguanosine. Serum malondialdehyde and glutathione levels were measured.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control (CONT): Obese patients who did not receive any drugs or herbal supplement were offered to be included in the CONT group.
- Orlistat (ORL): Obese patients who were treated with orlistat were offered to be included in the ORL group.
- Metformin (METF): Obese patients who were treated with metformin were offered to be included in the METF group.
- White Tea (WT): Obese patients who did not receive any drugs, but were taking white tea were offered to be included in the WT group.

SUMMARY:
Obesity is an increasing global public health issue. In general, tea consumption have been shown to offer benefit to obese patients. However, the potential of white tea (WT) to treat and protect from the adverse effects of obesity have not been addressed so far. The aim of this study was to examine the efficacy and impact WT consumption highest in catechins on levels of anthropometric and biochemical values in obese patients.

DETAILED DESCRIPTION:
Obesity is the increase in body weight above the normal level as a result of excessive fat accumulation. This condition is a chronic metabolic disease that increases the risk of long-term medical complications. The prevalence of obesity is an increasing global public health problem. Numerous conditions such as excessive and malnutrition, lack of physical activity, hormonal factors, genetic and psychological factors, and medicine use are effective in the formation of obesity. Obesity is associated with many diseases such as cardiovascular diseases, type 2 diabetes, hypertension, and dyslipidemia.

Since the mechanical load and myocardial metabolism increase in obesity, oxygen consumption also increases. Therefore, there is an increase in the formation of oxygen radicals (ROS) caused by mitochondrial respiration. Oxidative stress and ROS stimulate pro-inflammatory cytokine release. ROS attack macromolecules such as DNA, proteins, lipids. Macromolecular damage results in cellular damage and death. Damages caused by ROS are repaired by antioxidant defense systems. It has been suggested that inflammatory markers such as ghrelin, leptin, adiponectin, interleukins, matrix metalloproteinases, tumor necrosis factor are associated with insulin resistance in obese patients. These substances are effective on food intake, energy balance, insulin activity, lipid and glucose metabolism, angiogenesis and vascular structuring and blood pressure in the body.

Many drugs have been used to treat obesity. Orlistat is a widely used drug to treat this disease. It reversibly inhibits gastric and pancreatic lipases. Inactivation of lipases prevents the hydrolysis of triglycerides. Metformin, a dimethylbiguanide, inhibits the mitochondrial complex-I, which leads to adenosine 5-monophosphate activated protein kinase (AMPK) activation. By affecting the AMPK level, it provides the translocation of the glucose transporter 4 protein independently of insulin and regulates the blood glucose level. Clinicians often prescribe it to achieve weight loss. However, they have evinced serious adverse effects, including headache, cardiovascular diseases and depression, which restrict their use.

In recent years, one of the fastest growing fields in the treatment of obesity is the use of natural herbal products and many studies have proven the use of herbal products to be effective and safe. Especially, tea is reported to have anti-obesity, anti-diabetes, anti-inflammatory and hypolipidaemic actions.

Tea is produced from the leaves of the Camellia sinensis plant, which belongs to the Theaceae family, and is one of the most consumed beverages after water in many societies. In general, four types of tea are produced from the tea plant. WT differs from other teas in that only the buds and young leaves of the plant are used. WT has important benefits for human health with its high content of catechins and derivatives, as well as other tea components.

In the literature searches, no clinical research has been found on the effect of WT on obesity, which is richer than other tea varieties in terms of antioxidant properties and produced with less processing. This study aimed to determine the effect of WT consumption on obesity and the relationship between anthropometric and biochemical values of WT consumption in obese individuals.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index of 30 and above (kg/m²)

Exclusion Criteria:

* smoking
* physical disability preventing participating in the exercise programs
* joint problem preventing participating in the exercise programs
* trauma preventing participating in the exercise programs
* malignancy
* history of cerebrovascular disease
* active use of antidepressant drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese individuals who applied to the Endocrinology and Metabolism outpatient clinic of tertiary hospital.
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Weight loss | 3 months
  Decrease in body weight
Waist Circumference | 3 months
  Decrease in waist circumference
Body Mass Index | 3 months
  Decrease in body mass index

SECONDARY OUTCOMES:
Tumor Necrosis Factor - alpha | 3 months
  Decrease in serum Tumor Necrosis Factor - alpha level
Total cholesterol | 3 months
  Decrease in serum total cholesterol level
Low-Density Lipoprotein cholesterol | 3 months
  Decrease in serum Low-Density Lipoprotein cholesterol level
High-Density Lipoprotein cholesterol | 3 months
  Increase in serum High-Density Lipoprotein cholesterol level

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Yılmaz, Prof., Study Director — Recep Tayyip Erdogan University Medical Faculty
Locations (1):
- Recep Tayyip Erdogan University, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Sharing of individual participant data is prohibited by the Ethics committee. It is allowed on an individual basis.

REFERENCES:
- [Background] Castro-Barquero S, Lamuela-Raventos RM, Domenech M, Estruch R. Relationship between Mediterranean Dietary Polyphenol Intake and Obesity. Nutrients. 2018 Oct 17;10(10):1523. doi: 10.3390/nu10101523. PMID 30336572
- [Background] Taylor EB. The complex role of adipokines in obesity, inflammation, and autoimmunity. Clin Sci (Lond). 2021 Mar 26;135(6):731-752. doi: 10.1042/CS20200895. PMID 33729498
- [Background] Xia X, Lin Z, Shao K, Wang X, Xu J, Zhai H, Wang H, Xu W, Zhao Y. Combination of white tea and peppermint demonstrated synergistic antibacterial and anti-inflammatory activities. J Sci Food Agric. 2021 Apr;101(6):2500-2510. doi: 10.1002/jsfa.10876. Epub 2020 Oct 30. PMID 33058206
- [Background] Yang CS, Zhang J, Zhang L, Huang J, Wang Y. Mechanisms of body weight reduction and metabolic syndrome alleviation by tea. Mol Nutr Food Res. 2016 Jan;60(1):160-74. doi: 10.1002/mnfr.201500428. Epub 2015 Dec 9. PMID 26577614